CLINICAL TRIAL: NCT04301882
Title: An Observational Cohort Study of Clinical Outcomes After Antiviral Treatment of Chronic Hepatitis C Patients
Brief Title: An Observational Cohort Study of Clinical Outcomes After Antiviral Treatment of Chronic Hepatitis C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Director of Hepatology Division 2, Beijing Ditan Hospital
Other Study IDs: DTXY023
Record Dates: First submitted 2020-03-05; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Interferon; Ribavirin; Clinical outcome
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 144 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- interferon combined with ribavirin (PR) antiviral therapy: Patients with chronic hepatitis C treated with interferon combined with ribavirin (PR) antiviral therapy (PR therapy greater than or equal to 6 months)
  Interventions: Drug: interferon combined with ribavirin (PR) antiviral therapy
- direct antiviral drugs (DAAs): Patients with chronic hepatitis C treated with direct antiviral drugs (DAAs)
  Interventions: Drug: direct antiviral drugs (DAAs)

INTERVENTIONS:
Drug: interferon combined with ribavirin (PR) antiviral therapy — Patients with chronic hepatitis C treated with interferon combined with ribavirin (PR) antiviral therapy (PR therapy greater than or equal to 6 months)
  Groups: interferon combined with ribavirin (PR) antiviral therapy
Drug: direct antiviral drugs (DAAs) — Patients with chronic hepatitis C treated with direct antiviral drugs (DAAs)
  Groups: direct antiviral drugs (DAAs)

SUMMARY:
This study is a two-way, non-interventional long-term dynamic follow-up clinical observational cohort study. In the Second Division of Liver Diseases, Beijing Ditan Hospital, Capital Medical University, chronic hepatitis C patients who were treated with interferon combined with ribavirin (PR) antiviral therapy (PR treatment for 6 months or more) and / or direct acting antivirals (DAAs ), and the baseline, antiviral treatment and discontinuation follow-up data of patients before antiviral treatment were collected, and follow-up observations of patients were carried out for every 3-6 months. The clinical data such as clinical biochemistry, HCV RNA and serological indicators (anti-HCV), AFP, and liver imaging (liver ultrasound) were collected during the study period. The virological response and clinical outcomes of chronic hepatitis C antiviral therapy were observed for at least 144 weeks. The incidence of liver cancer and decompensated liver cirrhosis after discontinuation of the drug was the main evaluation index. The aim is to explore long-term virological response and clinical outcomes, and elucidate its influencing factors.

DETAILED DESCRIPTION:
This study is a two-way, non-interventional long-term dynamic follow-up clinical observational cohort study. Enrolled in the Second Division of Liver Diseases, Beijing Ditan Hospital, Capital Medical University, via interferon combined with ribavirin (PR) antiviral therapy (PR treatment for 6 months or more) and / or direct acting antivirals (DAAs ) For patients with chronic hepatitis C treated, collect baseline, antiviral treatment and discontinuation follow-up data of patients before antiviral treatment, and follow-up observations of patients enrolled every 3-6 months. Collect clinical data such as clinical biochemistry, HCV RNA and serological indicators (anti-HCV), AFP, and liver imaging (liver ultrasound) during the study period. The virological response and clinical outcomes of chronic hepatitis C antiviral therapy were observed for at least 144 weeks. The incidence of liver cancer and decompensated liver cirrhosis after discontinuation of the drug was the main evaluation index. The aim is to explore long-term virological response and clinical outcomes, and elucidate its influencing factors.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 75;
* Unlimited gender;
* Patients with chronic hepatitis C treated with interferon combined with ribavirin (PR) antiviral therapy (PR therapy for 6 months or more) and / or direct antiviral drugs (DAAs). All patients with chronic hepatitis C met the diagnostic criteria of the Chinese Guidelines for the Prevention and Treatment of Chronic Hepatitis C (2015)
* No hormones and / or immunosuppressants and other hepatoprotective drugs;
* Sign a written informed consent.

Exclusion Criteria:

* Combined with other hepatitis virus (HBV, HDV) infections;
* Immune liver disease;
* HIV infection;
* long-term alcohol and / or other liver damage drugs;
* mental illness;
* Evidence of liver tumor (liver cancer or AFP> 100 ng / ml);
* Decompensated cirrhosis;
* Those who have serious heart, brain, lung, kidney and other system diseases that cannot participate in long-term follow-up;
* There are hormones and / or immunosuppressants and other hepatoprotective drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C treated with interferon combined with ribavirin (PR) antiviral therapy (PR therapy for 6 months or more) and / or direct antiviral drugs (DAAs). All patients with chronic hepatitis C met the diagnostic criteria of the Chinese Guidelines for the Prevention and Treatment of Chronic Hepatitis C (2015).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of liver cancer | 144 weeks after withdrawal
  Incidence of liver cancer after chronic hepatitis C antiviral treatment
Incidence of decompensated cirrhosis | 144 weeks after withdrawal
  Incidence of decompensated cirrhosis after chronic hepatitis C antiviral treatment

SECONDARY OUTCOMES:
Rate of sustained virological response or relapse | 144 weeks after withdrawal
  Rate of sustained virological response or relapse after antiviral treatment of chronic hepatitis C

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatology Division 2, Beijing Ditan Hospital, Beijing, Beijing Municipality, China